CLINICAL TRIAL: NCT00439712
Title: Efficacy of Levocetirizine in the Treatment of Nasal Obstruction Due to Perennial Rhinitis
Brief Title: Levocetirizine in the Treatment of Nasal Obstruction Due to Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut für Atemwegsforschung GmbH (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Claus Bachert MD PhD, Institut für Atemwegsforschung GmbH
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Levo-6-06
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Experimental)
  Interventions: Drug: Levocetirizine
- Treatment Group 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levocetirizine — 1 tablet of Levocetirizine 5 mg OD in the morning for 29+/-4 days
  Arms: Treatment Group 1
Drug: Placebo — 1 placebo tablet OD in the morning for 29+/-4 days
  Arms: Treatment Group 2

SUMMARY:
The purpose of this study is to show that in patients suffering from perennial allergic rhinitis levocetirizine 5 mg OD relieves nasal obstruction. Furthermore the study is to investigate how relevant for these patients their nasal obstruction and the effect of levocetirizine on their nasal obstruction are.

DETAILED DESCRIPTION:
The study is performed according to a monocentre, double-blind, placebo controlled, two arm parallel group design. It is divided in 3 periods: A 7 ± 2 day screening phase when patients are not to treat their perennial allergic rhinitis (PAR) is followed by a 29 ± 4 day treatment period when patients administer either levocetirizine 5 mg OD or placebo and a 14 ± 2 week post treatment observation period when again medication against PAR is not to be taken. However in all study periods patients are provided cromoglicine nasal spray and eye drops which in case of severe complaints they may use as rescue medication.

Throughout the study patients keep a diary documenting the severity of their nasal and ocular symptoms of allergy. Every morning and every evening they use a 4-point scale (0 = no symptom, 1 = mild, 2 = moderate, 3 = severe) to rate nasal obstruction, rhinorrhea, nasal itching, sneezing and ocular complaints they experienced during the preceding 12 hours. Furthermore they report adverse events and intake of drugs inclusive of rescue and (during treatment period) study medication.

Patients attend 5 visits to the study site. On visit 1 medical history and concomitant medication are assessed and patients undergo a physical examination, a pregnancy test in case of women of child bearing potential, and, if necessary, a skin prick test. Blood is taken to estimate creatinine clearance. Inclusion and exclusion criteria are checked and, if they do not contradict study continuation, patients enter the screening period which ends in the morning of the day visit 2. If on this visit morning diary reports show sufficiently high nasal obstruction scores and study participation still complies with the inclusion and exclusion criteria, patients are randomized and start the treatment period taking the first dose at the study site. On visit 2 as well as on the following visits adverse events and use of medication are surveyed and compliance is checked. Visit 3, 4 and 5 are scheduled after one week of treatment, between treatment and post treatment observation period and at the end of the study respectively. On visit 5 there is a final physical examination and again females of childbearing potential undergo a pregnancy test. To assess how relevant for patients nasal obstruction and the effect of the study medication on nasal obstruction are questionnaires are completed on each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 to 65 years (inclusively).
* Ability to understand nature, scope and possible consequences of the study.
* Capability and willingness to comply with the requirements of the protocol.
* Written informed consent was granted after in depth written and oral information on all relevant aspects of the study.
* Adequate contraception in case of females of child bearing potential (i.e. hormonal contraception, IUD, double barrier method, monogamous sexual relation with an monogamous partner, sexual inactivity).
* At least 2 year history of perennial allergic rhinitis with pronounced symptoms.
* Sensitization to D. farinae or D. pteronyssinus proved by a prick test (wheal diameter ≥ 3 mm) or measurement of specific IgE (at least RAST class 2) at most one year ago.
* On visit 2: Sum of the morning nasal obstruction scores documented in the screening diary is at least 40% of the maximal sum the patient could have attained.

Exclusion Criteria:

* Exposure to another investigational agent within the last three months.
* Pregnancy or nursing.
* Severe diseases and diseases, conditions or findings which might interfere with the study results, deteriorate due to study participation or require impermissible medication. In particular this includes

  * restricted liver or kidney function or respectively creatinine clearance below 50 ml/min, the clearance being estimated according to the formula by Cockcroft/Gault from serum creatinine assessed on visit 1,
  * nasal polyps, severe deviations of the nasal septum, and any other considerable impairments of nasal patency,
  * an ear, nose or throat infection during the last 2 weeks or any other but allergic form of rhinitis,
  * asthma requiring any other treatment than short acting β-agonists on demand,
  * atopic dermatitis with considerable probability to require corticosteroid treatment.
* Intake of impermissible medication or non observance of the designated washout periods.
* History of malignancy within the last 5 years.
* Drug or alcohol abuse.
* Intention to donate blood during the study period.
* Intolerance to one of the components of the trial medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Average morning nasal obstruction score calculated from diary assessments during treatment. | 4 week treatment period

SECONDARY OUTCOMES:
average morning and average evening single symptom score calculated from diary assessments during treatment period (with exception of the primary endpoint) | 4 week treatment period
average of the daily mean single symptom score (mean of morning and evening assessment) calculated with respect to diary assessments during treatment period | 4 week treatment period
average morning, evening and total T5SS calculated with respect to the treatment period | 4 week treatment period
average use of rescue medication (number of applications) during the treatment period | 4 week treatment period
differences between the preceding parameters and the respective averages calculated in regard to the follow-up period | 4 week treatment and 2 week follow-up period
results and changes in results of questionnaire 1 | assessed on visits during the 7 week study period
results of questionnaires 2, 3 and 4 | assessed on visits during the 4 week treatment and the 2 week follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bachert, MD, PhD, Principal Investigator — Institut für Atemwegsforschung GmbH
Locations (1):
- Institut für Atemwegsforschung GmbH, Düsseldorf, North Rhine-Westphalia, Germany